CLINICAL TRIAL: NCT02483156
Title: Randomized, Open-Label, Study to Evaluate the Safety and Efficacy of Sofosbuvir Tablet Plus Ribavirin Tablet (Part A) Versus Single Dose (2 Tablets) of EHCV Containing Sofosbuvir, Ribavirin, and Natural Anti-hemolytic (B) in Egyptian Adults With Chronic Genotype 4 HCV Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Egyptian Liver Hospital (Other)
Collaborators: Wadi El Nil Hospital (Unknown)
Responsible Party: Principal Investigator, Dr.Waleed Samir, Director of Clinical and Research Laboratory & Head of Molecular Biology Unit., Egyptian Liver Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELH - 2015
Record Dates: First submitted 2015-06-19; First posted 2015-06-26 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Hepatitis c
Keywords: HCV; Sofosbuvir; Ribavirin
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin; Sofosbuvir

ARMS (2):
- SOF + RBV (Active Comparator): Sofosbuvir 400 mg once daily +RBV (1000 mg/day) for 12-24 weeks
  Interventions: Drug: Sofosbuvir tablet (SOF) 400 mg - once daily; Drug: Ribavirin (RBV) 1000 mg - splitted on 2 doses daily - 600 mg on morning and 400 mg on evening
- sof + RBV + AH (Experimental): Single Dose (2 tablets) once daily each tablet containing SOF 200 mg, RBV 500 mg and Natural anti-hemolytic (AH) at 200 mg for 12-24 weeks
  Interventions: Drug: Two tablets of EHCV in Single Dose each tablet containing SOF 200 mg, RBV 500 mg and Natural anti-hemolytic (AH) at 200 mg

INTERVENTIONS:
Drug: Two tablets of EHCV in Single Dose each tablet containing SOF 200 mg, RBV 500 mg and Natural anti-hemolytic (AH) at 200 mg — The fixed dose EHCV combinations in Single Dose (2 tablets) once daily each tablet containing SOF 200 mg, RBV 500 mg, and Natural anti-hemolytic (AH) at 200 mg. Subjects will take 2 tablet with food for 12-24 weeks.
  Arms: sof + RBV + AH
Drug: Sofosbuvir tablet (SOF) 400 mg - once daily — SOF is manufactured as a 400 mg tablet for oral administration. Subjects will take 1 tablet for a total dose of 400 mg orally once daily in the morning with RBV and with food for 12-24 weeks.
  Arms: SOF + RBV
Drug: Ribavirin (RBV) 1000 mg - splitted on 2 doses daily - 600 mg on morning and 400 mg on evening — RBV (1000 mg.) splitted on 2 doses daily - 600 mg on morning and 400 mg on evening with SOF and with food for 12-24 weeks.
  Arms: SOF + RBV

SUMMARY:
Two Groups of Genotype 4 HCV Patients will participate through open-label randomized Study comparing Sofosbuvir tablet Plus Ribavirin tablet (Part A) versus single Dose (2 tablets) of EHCV containing Sofosbuvir, Ribavirin, and Natural anti-hemolytic (B) evaluating the safety and efficacy for both arms.

Sponsor: Wadi El Nil Hospital

Study Centers Planned: Approximately 2 sites in Egypt

DETAILED DESCRIPTION:
Study Design:

Part A

Randomized, open-label study in treatment naïve and treatment experienced adults with chronic genotype 4 HCV infection.

Treatment-naïve is defined as having never received treatment for HCV with any interferon (IFN), RBV, or other approved or experimental HCV specific direct acting antivirals.

Treatment-experienced is defined as:

1. IFN Intolerant
2. Non-response
3. Relapse/Breakthrough

It is planned that 40 + 40 subjects will be enrolled in the study such that an approximate even number of treatment naïve and treatment experienced subjects will be enrolled across the 2 treatment arms:

Arm 1 Sofosbuvir 400 mg once daily +RBV (1000 mg/day) for 12-24 weeks

Arm 2 Single Dose (2 tablets) once daily each tablet containing SOF 200 mg, RBV 500 mg, and Natural anti-hemolytic (AH) at 200 mg for 12-24 weeks Treatment assignments will be stratified according to prior treatment experience and the presence or absence of cirrhosis.

Cohorts:

Cohort is a single-arm, open-label, non-randomized design in subjects who completed treatment in Part A of the study with SOF+RBV for 12-24 weeks or in Part B of the study with single dose EHCV (2 Tablet) containing SOF/RBV/AH FDC for 12-24 weeks.

Diagnosis and Main Eligibility Criteria: HCV RNA > 104 IU/mL or HCV RNA > LLOQ and did not achieve SVR 12 after completing prior treatment in this study with chronic genotype 4 HCV infection. Treatment-naïve or treatment experienced adults, male and non-pregnant/non-lactating female subjects, ages 18 years or older. See Section 1 and 1.2 of the protocol for detailed Inclusion and Exclusion criteria.

Study Procedures/

Frequency: Study visits for all subjects will occur at screening, Baseline/Day 1. On-treatment visits will occur as follows:

• Part A, Arm 1 and 2 - at the end of Weeks 1, 2, 4, 6, 8, 10, 12, 16, 20, and 24 All subjects will complete a 4-Week Post-treatment visit regardless of treatment duration. Subjects with HCV RNA < LLOQ will continue to 12 Week and 24 Week Post treatment visits unless confirmed viral relapse occurs at which time subjects will be early terminated from the study.

Screening assessments include safety laboratory tests (chemistry, hematology, coagulation, and urinalysis), 12 lead ECG, HCV RNA, serology (HBV, and HIV), hemoglobin A1c, urine drug screen, liver imaging, serum B-hCG (for all female subjects of child-bearing potential), physical examination (with height and bodyweight), vital signs, medical history, concomitant medications, and adverse events. In addition, subjects being screened for Part A and Part B (Cohort 1) will have HCV genotyping and IL28B genotyping performed.

On-treatment assessments include safety laboratory tests (chemistry, hematology, and coagulation), HCV RNA, urine pregnancy tests (for all female subjects of child-bearing potential), physical examination, vital signs, concomitant medications, and adverse events.

Post-treatment assessments include HCV RNA, urine pregnancy tests (for all female subjects of child-bearing potential), vital signs, concomitant medications, and adverse events.

Samples will be collected at Baseline/Day 1 and every visit Plasma samples will be collected during treatment visits for pharmacokinetic (PK) analysis of study drug (Part A only). Untested samples will be archived for up to 10 years.

Test Product, Dose, and Mode of Administration: SOF is manufactured as a 400 mg tablet for oral administration. Subjects will take 1 tablet for a total dose of 400 mg orally once daily in the morning with RBV (1000 mg) splitted on 2 doses daily 600 mg on morning and 400 mg on evening and with food for 12-24 weeks.

The fixed dose EHCV combinations in Single Dose (2 tablets) once daily each tablet containing SOF 200 mg, RBV 500 mg, and Natural anti-hemolytic (AH) at 200 mg. Subjects will take 2 tablet with food for 12-24 weeks.

Reference Therapy, Dose, and Mode of Administration: None

Criteria for Evaluation:

Safety: Adverse events will be collected from baseline through the 4 Week Post-Treatment Visit and AEs related to study procedures, will be collected from when subjects sign the consent form. Clinical laboratory tests will be performed during treatment through the 12 Week Post-Treatment Visit.

Efficacy: Efficacy will be evaluated using scheduled assessments of HCV RNA performed using COBAS® TaqMan® HCV Test, v2.0 for Use with the High Pure System.

PK Part A only. A single PK blood sample will be collected at all study visits while on Treatment.

Statistical Methods: The primary efficacy endpoint is SVR12 (ie, HCV RNA < LLOQ 12 weeks post-treatment) in all subjects who are randomized and treated. No statistical hypothesis testing will be performed. For each of the two treatment groups, a 2-sided 95% confidence interval using the exact binomial distribution will be constructed.

Part A: With a sample size of 40 subjects in each arm, a two sided 95% exact confidence interval will extend at most 29% in length.

Part B: With a sample size of 40 subjects in each treatment group in Cohort 1, a 2-sided 95% exact confidence interval will extend at most 32% in length.

Secondary efficacy endpoints include the proportion of subjects with SVR4 and SVR24.

All continuous endpoints will be summarized using an 8 number summary (n, mean, standard deviation, and median, Q1, Q3, minimum, maximum) by treatment duration. All categorical endpoints will be summarized by number and percentage of subjects who meet the endpoint definition.

Safety endpoints will be analyzed by the number and percent of subjects with events or abnormalities for categorical values or using an 8 number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum) for continuous data by treatment group.

Data from Part B will be analyzed separately from Part A and may be reported separately.

This study will be conducted in accordance with the guidelines of Good Clinical Practices (GCPs) including archiving of essential documents.

ELIGIBILITY:
Inclusion Criteria

Inclusion Criteria for Part A

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study.

1. Willing and able to provide written informed consent.
2. Male or female, age ≥ 18 years.
3. HCV RNA ≥ 104 IU/mL at screening.
4. Confirmed chronic HCV infection as documented by either:

   a. a positive anti-HCV antibody test or positive HCV RNA or positive HCV genotyping test at least 6 months prior to the Baseline/Day 1 visit, or
5. HCV genotype 4 at screening as determined by the Central Laboratory. Any non-definitive results will exclude the subject from study participation.
6. The subject's medical records must be sufficient to categorize prior treatment history as one of the following:

   i) IFN-intolerant: subject had documented intolerance to IFN during prior IFN therapy of up to 12 weeks duration ii) Non-response: subject did not achieve undetectable HCV RNA levels on treatment iii) Relapse/Breakthrough: subject achieved undetectable HCV RNA levels during treatment or within 4 weeks after treatment and later showed detectable HCV RNA

   An Absence of cirrhosis is defined as any one of the following:
   * Liver biopsy within 2 years of Screening showing absence of cirrhosis
   * Fibroscan with a result of ≤ 12.5 kPa within 6 months of Baseline/Day1
   * FibroTest score of ≤ 0.48 AND APRI of ≤ 1 performed during Screening In the absence of a definitive diagnosis of the presence or absence of cirrhosis by the above criteria, a liver biopsy is required. Liver biopsy results supersede the results obtained by Fibroscan or Fibro Test.
7. Body mass index (BMI) ≥ 18 kg/m2.
8. Screening ECG without clinically significant abnormalities.
9. Subjects must have the following laboratory parameters at screening:

   * ALT ≤ 10 x the upper limit of normal (ULN)
   * AST ≤ 10 x ULN
   * Hemoglobin ≥ 12 g/dL for male, ≥ 11 g/dL for female subjects
   * Platelets > 50,000 cells/mm3
   * INR ≤ 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR
   * Albumin ≥ 3 g/dL
   * Direct bilirubin ≤ 1.5 x ULN
   * HbA1c ≤ 10%
   * Creatinine clearance (CLcr) ≥ 60 mL/min, as calculated by the Cockcroft-Gault equation
10. Subject has not been treated with any investigational drug or device within 30 days of the screening visit.
11. A female subject is eligible to enter the study if it is confirmed that she is:

    1. Not pregnant or nursing
    2. Of non-childbearing potential (ie, women who have had a hysterectomy, both ovaries removed or medically documented ovarian failure, or are postmenopausal women > 50 years of age with cessation [for 12 months] of previously occurring menses), or
    3. Of childbearing potential (ie, women who have not had a hysterectomy, both ovaries removed, or no medically documented ovarian failure). Women ≤ 50 years of age with amenorrhea will be considered to be of childbearing potential. These women must have a negative serum pregnancy test at screening and a negative urine pregnancy test on the Baseline/Day 1 visit prior to randomization. They must also agree to one of the following from 3 weeks prior to Baseline/Day 1 until 6 months after last dose of RBV:

       * Complete abstinence from intercourse. Periodic abstinence from intercourse (eg, calendar, ovulation, symptothermal, post-ovulation methods) is not permitted.

    Or
    * Consistent and correct use of 1 of the following methods of birth control listed below in addition to a male partner who correctly uses a condom from the date of screening until 6 months after the last dose of RBV. Women of childbearing potential must not rely on hormone-containing contraceptives as a form of birth control during the study. Female subjects using a hormone-containing contraceptive prior to screening may continue their contraceptive regimen in addition to the study specified methods of birth control.
    * Intrauterine device (IUD) with a failure rate of < 1% per year
    * Female barrier method: cervical cap or diaphragm with spermicidal agent
    * Tubal sterilization
    * Vasectomy in male partner
12. All male study participants must agree to consistently and correctly use a condom, while their female partner agrees to use either 1 of the non-hormonal methods of birth control listed above or a hormone-containing contraceptive listed below, from the date of screening until 7 months after their last dose of RBV:

    * Implants of levonorgestrel
    * Injectable progesterone
    * Oral contraceptives (either combined or progesterone only)
    * Contraceptive vaginal ring
    * Transdermal contraceptive patch
13. Male subjects must agree to refrain from sperm donation for at least 7 months after the last dose of RBV.
14. Subject must be of generally good health as determined by the Investigator.
15. Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.

Inclusion Criteria for Part B

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study.

1. Willing and able to provide written informed consent.
2. Male or female, age ≥ 18 years.
3. HCV genotype 4 at screening as determined by the Central Laboratory. Any non-definitive results will exclude the subject from study participation. Historical result from prior participation in this study is acceptable, if applicable.
4. Cohort 1 only: HCV RNA ≥ 104 IU/mL at screening.
5. Chronic HCV infection (≥ 6 months) documented by medical history.
6. Cohort 1 only: HCV treatment naïve, defined as no prior exposure to any IFN, RBV, or other approved or experimental HCV specific direct acting antiviral agent
7. BMI ≥ 18 kg/m2

   Absence of cirrhosis is defined as any one of the following:
   1. Liver biopsy within 2 years of Screening showing absence of cirrhosis
   2. Fibroscan with a result of ≤ 12.5 kPa within 6 months of Baseline/Day1 C- Fibro Test score of ≤ 0.48 AND APRI of ≤ 1 performed during Screening

   In the absence of a definitive diagnosis of the presence or absence of cirrhosis by the above criteria, a liver biopsy is required. Liver biopsy results supersede the results obtained by Fibroscan or Fibro Test.
8. Screening ECG without clinically significant abnormalities.
9. Subjects must have the following laboratory parameters at screening:

   * ALT ≤ 10 x the upper limit of normal (ULN)
   * AST ≤ 10 x ULN
   * Hemoglobin ≥ 12 g/dL for male, ≥ 11 g/dL for female subjects
   * Platelets > 50,000 cells/mm3
   * INR ≤ 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR
   * Albumin ≥ 3 g/dL
   * Direct bilirubin ≤ 1.5 x ULN
   * HbA1c ≤ 10%
   * Creatinine clearance (CLcr) ≥ 60 mL/min, as calculated by the Cockcroft-Gault equation

   Subjects who received prior treatment in this study and who currently do not fulfill all of the above requirements may be enrolled in Part B Cohort 2 at the request of the Investigator and with the approval of the Medical Monitor or Study Director.
10. Subject has not been treated with any investigational drug or device within 28 days of the Baseline/Day 1 visit.
11. A female subject is eligible to enter the study if it is confirmed that she is:

    D Not pregnant or nursing e Of non-childbearing potential (ie, women who have had a hysterectomy, both ovaries removed or medically documented ovarian failure, or are postmenopausal women > 50 years of age with cessation [for 12 months] of previously occurring menses), or

    F Of childbearing potential (ie, women who have not had a hysterectomy, both ovaries removed, or no medically documented ovarian failure). Women ≤ 50 years of age with amenorrhea will be considered to be of childbearing potential. These women must have a negative serum pregnancy test at screening and a negative urine pregnancy test on the Baseline/Day 1 visit prior to randomization. They must also agree to one of the following from 3 weeks prior to Baseline/Day 1 until 30 days after the last dose of LDV/SOF or 6 months after last dose of RBV:

    • Complete abstinence from intercourse. Periodic abstinence from intercourse (eg, calendar, ovulation, symptothermal, post-ovulation methods) is not permitted.

    Or
    * Consistent and correct use of 1 of the following methods of birth control listed below in addition to a male partner who correctly uses a condom from the date of screening until 30 days after the last dose of LDV/SOF or 6 months after the last dose of RBV.
    * Intrauterine device (IUD) with a failure rate of < 1% per year
    * Female barrier method: cervical cap or diaphragm with spermicidal agent
    * Tubal sterilization
    * Vasectomy in male partner
    * Implants of levonorgestrel
    * Injectable progesterone
    * Oral contraceptives (either combined or progesterone only)
    * Contraceptive vaginal ring
    * Transdermal contraceptive patch
12. All male study participants must agree to consistently and correctly use a condom from Baseline until 90 days after their last dose of LDV/SOF or 7 months after their last dose of RBV. If their female partner is of childbearing potential (as defined above), she must use 1 of the methods of birth control listed above from the date of screening until 90 days after their last dose of LDV/SOF or 7 months after their last dose of RBV.
13. Male subjects must agree to refrain from sperm donation for at least 7 months after the last dose of RBV or 90 days after their last dose of LDV/SOF, as applicable.
14. Subject must be of generally good health as determined by the Investigator.
15. Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.

Exclusion Criteria

Exclusion Criteria for Part A

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

1. for treatment naïve subjects only: Prior exposure to IFN, RBV, or other approved or experimental direct-acting antiviral targeting the HCV.
2. for treatment-experienced subjects: prior exposure to a NS5a inhibitor, NS5b nucleotide inhibitor, or NS5b non-nucleotide inhibitor targeting the HCV
3. Pregnant or nursing female or male with pregnant female partner.
4. Chronic liver disease of a non-HCV etiology (eg, hemochromatosis, Wilson's disease, α1 antitrypsin deficiency, cholangitis).
5. Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV).
6. Contraindication to RBV therapy e.g., history of clinically significant hemoglobinopathy (sickle cell disease, thalassemia).
7. History of malignancy diagnosed or treated within 5 years (recent localized treatment of squamous or non-invasive basal cell skin cancers is permitted; cervical carcinoma in situ is allowed if appropriately treated prior to screening); subjects under evaluation for malignancy are not eligible.
8. Chronic use of systemically administered immunosuppressive agents (eg, prednisone equivalent > 10 mg/day).
9. Clinically-relevant drug or alcohol abuse within 12 months of screening. A positive drug screen will exclude subjects unless it can be explained by a prescribed medication; the diagnosis and prescription should be approved by the investigator.
10. History of solid organ transplantation.
11. Current or prior history of clinical hepatic decompensation (eg, ascites, variceal hemorrhage, hepatic encephalopathy, hepatorenal syndrome and hepatopulmonary syndrome).
12. History of clinically-significant illness or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol.
13. History of a gastrointestinal disorder (or post-operative condition) that could interfere with the absorption of the study drug.
14. History of significant pulmonary disease, significant cardiac disease or porphyria.
15. Excessive alcohol ingestion, defined as 3 glasses/day (1 glass is equivalent to 284 mL beer, 125 mL wine, or 25 mL distilled spirits) for females and 4 glasses/day for males.
16. History of difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
17. Donation or loss of more than 400 mL blood within 2 months prior to Baseline/Day 1.
18. Known hypersensitivity to RBV, the study investigational medicinal product, the metabolites, or formulation excipients.

Exclusion Criteria for Part B

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

1. For treatment naïve subjects only (Cohort 1): Prior exposure to IFN, RBV, or other approved or experimental direct-acting antiviral targeting the HCV.
2. Current or prior history of any of the following:

   A Clinical hepatic decompensation (ie, ascites, encephalopathy or variceal hemorrhage) B Clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol, or, current evaluation for a potentially clinically significant illness (other than HCV) C Gastrointestinal disorder or post-operative condition that could interfere with the absorption of the study drug D Solid organ transplantation E Significant pulmonary disease, significant cardiac disease or porphyria F Psychiatric hospitalization, suicide attempt, and/or a period of disability as a result of their psychiatric illness within the last 5 years Subjects with psychiatric illness (without the prior mentioned conditions) that is well-controlled on a stable treatment regimen for at least 6 months prior to Baseline/Day 1 or that has not required medication in the last 12 months may be enrolled.

   G Any malignancy within the 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc.), or current evaluation for possible malignancy H Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy I Significant drug allergy (such as anaphylaxis or hepatotoxicity)
3. Chronic liver disease of a non-HCV etiology (eg, hemochromatosis, Wilson's disease, α1 antitrypsin deficiency, cholangitis)
4. Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
5. Use of any prohibited concomitant medications
6. Contraindication to RBV therapy, including significant history of clinically significant hemoglobinopathy (eg, sickle cell disease, thalassemia)
7. In the judgment of the investigatory, any clinically-relevant drug or alcohol abuse within 12 months of screening that may interfere with subject treatment, assessment of compliance with the protocol
8. Pregnant or nursing females or male with pregnant female partner
9. Known hypersensitivity to RBV, SOF, or formulation excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Experienced Adverse Events During Treatment Period | Baseline to 4 Week Post-Treatment Visit
  Adverse events will be collected from baseline through the 4 Week Post-Treatment Visit and AEs related to study procedures, will be collected from when subjects sign the consent form.

SECONDARY OUTCOMES:
Change in Circulating HCV RNA | Baseline to 24 weeks after discontinuation of therapy
  Efficacy will be evaluated using scheduled assessments of HCV RNA performed using COBAS® TaqMan® HCV Test, v2.0 for Use with the High Pure System.

OTHER OUTCOMES:
Change in the circulating Non-genetic biomarkers | Baseline to 24 week ( treatment period)
  To explore the utility of non-genetic biomarkers, such as IP10, in predicting the natural history of disease, virologic response to therapy, and/or the tolerability of medical therapies

CONTACTS AND LOCATIONS:
Locations (1):
- Egyptian Liver Hospital, Sherbin, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Doss W, Shiha G, Hassany M, Soliman R, Fouad R, Khairy M, Samir W, Hammad R, Kersey K, Jiang D, Doehle B, Knox SJ, Massetto B, McHutchison JG, Esmat G. Sofosbuvir plus ribavirin for treating Egyptian patients with hepatitis C genotype 4. J Hepatol. 2015 Sep;63(3):581-5. doi: 10.1016/j.jhep.2015.04.023. Epub 2015 May 1. PMID 25937436
- [Derived] Shiha G, Soliman R, Elbasiony M, Darwish NHE, Mousa SA. Novel combined single dose anti-hepatitis C therapy: a pilot study. Sci Rep. 2021 Feb 25;11(1):4623. doi: 10.1038/s41598-021-84066-3. PMID 33633233
- See also: Egyptian Liver Hospital site — http://www2.mans.edu.eg/hosted/liver-ri/en/about_institute.htm